CLINICAL TRIAL: NCT03428828
Title: Amygdala rtfMRI Neurofeedback for Treatment Resistant Depression
Brief Title: Neurofeedback for Treatment Resistant Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kymberly Young (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Kymberly Young, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY19020313; R61MH115927 (NIH)
Record Dates: First submitted 2018-02-01; First posted 2018-02-12 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Treatment Resistant Depression
Keywords: Neurofeedback; major depressive disorder; treatment resistant; amygdala
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Amygdala Neurofeedback (Experimental): attempt to up regulate the left amygdala during positive autobiographical memory recall via real time fMRI neurofeedback from the amygdala. Five sessions will be performed within a 2 month period.
  Interventions: Device: Amygdala Neurofeedback
- Parietal Neurofeedback (Active Comparator): attempt to upregulate the left horizontal segment of the intraparietal sulcus, a region not involved in emotional processing, during positive autobiographical memory recall via real time fMRI neurofeedback. Five sessions will be performed within a 2 month period.
  Interventions: Device: Parietal Neurofeedback

INTERVENTIONS:
Device: Amygdala Neurofeedback — Participants are shown activity from their left amygdala in real time and are instructed to increase the level of activity in that region by thinking of positive autobiographical memories
  Arms: Amygdala Neurofeedback
Device: Parietal Neurofeedback — Participants are shown activity from their left horizontal segment of the intraparietal sulcus in real time and are instructed to increase the level of activity in that region by thinking of positive autobiographical memories
  Arms: Parietal Neurofeedback

SUMMARY:
The purpose of this study is to determine the clinical efficacy of real-time functional magnetic resonance imaging neurofeedback (rtfMRI-nf) training to increase the amygdala's response to positive autobiographical memories in patients with depression who are considered treatment-resistant

DETAILED DESCRIPTION:
Up to two-thirds of patients diagnosed with major depressive disorder (MDD) will not respond to standard pharmacological and psychological interventions and will be considered treatment resistant (TR-MDD). Decreased reactivity to positive stimuli, indexed by low amygdala reactivity to positive autobiographical memory recall, may be a causal mechanism interfering with recovery from TR-MDD. Previous work in our lab suggests that individuals who do respond to antidepressant medications show increased amygdala activity that is indistinguishable from controls relative to baseline, while TR-MDD individuals fail to show this increase in amygdala activity. Furthermore, the investigators have found that MDD participants (more generally, not specifically TR- MDD) are indeed able to increase their amygdala response during positive memory recall via real-time fMRI neurofeedback (rtfMRI-nf) training, and that this increase is associated with large and rapid reductions in depressive symptoms. Here, the investigators propose to evaluate whether rtfMRI-nf training to increase the amygdala response to positive memories may serve as an intervention for TR-MDD. 100 TR-MDD individuals will be randomly assigned under double-blind conditions to receive 5 amygdala rtfMRI-nf or 5 control rtfMRI-nf sessions where they are trained to regulate a parietal region putatively not involved in emotional processing or MDD. The investigators will assess changes in amygdala activity, severity of clinical symptoms, and autobiographical memory deficits. Success will suggest a new non- pharmacological, non-invasive intervention for a traditionally treatment-resistant population of MDD individuals.

ELIGIBILITY:
Inclusion Criteria:

* right-handed adults (ages 18 - 55) with a primary diagnosis of MDD according to diagnostic criteria DSM-5 for recurrent MDD who are currently depressed will be recruited to participate
* must be able to give written informed consent prior to participation
* must have fewer than 45% memories categorized as specific on the Autobiographical Memory Test
* must have a SHAPS score > 4, indicating the presence of anhedonia
* unmedicated or stable on an SSRI antidepressant regime (at least 3 weeks to ensure symptoms are stable)
* previously failed to respond to two previous SSRI medications according to either a medical record review or clinical interview during Visit 1

Exclusion Criteria:

* have a clinically significant or unstable cardiovascular, pulmonary, endocrine, neurological, gastrointestinal illness or unstable medical disorder
* met DSM-IV criteria for alcohol and/or substance dependence (other than nicotine) within 12 months prior to screening
* have a history of traumatic brain injury
* are unable to complete MRI scan due to claustrophobia or general MRI exclusions (e.g., shrapnel inside body)
* are currently pregnant or breast feeding
* are unable to complete questionnaires written in English
* current (within 3 weeks of testing) use of any antipsychotics, anticonvulsants, stimulants, benzodiazepines, beta-blockers, or other medications (except SSRI antidepressants) likely to influence cerebral blood flow. Effective medications will not be discontinued for the purposes of the study. Inclusion of patients on stable antidepressant medications was decided in order to allow generalization towards a real world population
* have a DSM-5 diagnosis of psychotic or organic mental disorder, bipolar I or II disorder or any past or current manic or hypomanic symptoms, autism, or a primary diagnosis of an anxiety disorder (though co-morbid anxiety will not be excluded)
* have any eye problems or difficulties in corrected vision.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-22 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory (BDI-II) | 12 weeks

SECONDARY OUTCOMES:
Amygdala Activity | 8 weeks
  % signal change from initial baseline to final transfer run in amygdala activity during ftMRI-nf sessions

CONTACTS AND LOCATIONS:
Overall Officials: Kymberly Young, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
The final data set will include self-reported demographic and behavioral data, clinical-rated information regarding illness course, severity, and comorbidities, and brain-imaging data collected during fMRI. The dataset will be stripped of identifiers prior to release for sharing, and will be shared openly and timely in accordance with the most recent NIH guidelines. Data will be shared every six months on the NIH-supported National Database for Clinical Trials Related to Mental Illness (NDCT) data repository.

REFERENCES:
- [Background] Young KD, Siegle GJ, Zotev V, Phillips R, Misaki M, Yuan H, Drevets WC, Bodurka J. Randomized Clinical Trial of Real-Time fMRI Amygdala Neurofeedback for Major Depressive Disorder: Effects on Symptoms and Autobiographical Memory Recall. Am J Psychiatry. 2017 Aug 1;174(8):748-755. doi: 10.1176/appi.ajp.2017.16060637. Epub 2017 Apr 14. PMID 28407727
- [Derived] Compere L, Siegle GJ, Lazzaro S, Riley E, Strege M, Canovali G, Barb S, Huppert T, Young K. Amygdala real-time fMRI neurofeedback upregulation in treatment resistant depression: Proof of concept and dose determination. Behav Res Ther. 2024 May;176:104523. doi: 10.1016/j.brat.2024.104523. Epub 2024 Mar 15. PMID 38513424